CLINICAL TRIAL: NCT02243371
Title: A Randomized Phase 2 Study of the Safety, Efficacy, and Immune Response of GVAX Pancreas Vaccine (With Cyclophosphamide) and CRS-207 With or Without Nivolumab in Patients With Previously Treated Metastatic Pancreatic Adenocarcinoma
Brief Title: GVAX Pancreas Vaccine (With CY) and CRS-207 With or Without Nivolumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry); Stand Up To Cancer (Other); Aduro Biotech, Inc. (Industry); American Association for Cancer Research (Other); Lustgarten Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J14113; ADU-CL-06; IRB00043936 (Other: JHMIRB)
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-02

CONDITIONS: Previously Treated Metastatic Adenocarcinoma of the Pancreas
MeSH Terms: interventions — Nivolumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: CY/ GVAX/ CRS-207/ nivolumab (Experimental)
  Interventions: Biological: CRS-207; Drug: nivolumab; Biological: GVAX; Drug: CY
- Arm B: CY/ GVAX/ CRS-207 (Experimental)
  Interventions: Biological: CRS-207; Biological: GVAX; Drug: CY

INTERVENTIONS:
Biological: CRS-207 — 1 × 10^9 CFU administered IV on Day 2 of Cycles 3-6
  Arms: Arm A: CY/ GVAX/ CRS-207/ nivolumab
Biological: CRS-207 — 1 × 10^9 CFU administered IV on Day 1 of Cycles 3-6
  Arms: Arm B: CY/ GVAX/ CRS-207
Drug: nivolumab — 3 mg/kg administered IV on Day 1 of Cycles 1-6
  Other Names: BMS-936558; anti-PD-1 mAb
  Arms: Arm A: CY/ GVAX/ CRS-207/ nivolumab
Biological: GVAX — 5x10^8 cells administered in 6 intradermal injections on Day 2 of Cycles 1 and 2
  Other Names: GVAX pancreas vaccine, Panc 10.05 pcDNA-1/GM-Neo, Panc 6.03 pcDNA-1/GM-Neo
Drug: CY — 200 mg/m^2 administered IV on Day 1 of Cycles 1 and 2
  Other Names: Cytoxan, Cyclophosphamide

SUMMARY:
The primary objective of this study is to compare the overall survival (OS) of subjects with previously treated metastatic pancreatic cancer treated with cyclophosphamide (CY)/nivolumab/GVAX pancreas vaccine followed by nivolumab/CRS-207 (Arm A) to subjects treated with CY/GVAX pancreas vaccine followed by CRS-207 (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Have histologically- or cytologically-proven adenocarcinoma of the pancreas. Patients with mixed histology will be excluded.
* Have metastatic disease.
* Have failed only 1 prior chemotherapy regimen for metastatic pancreatic cancer.
* Patients with the presence of at least one measurable lesion.
* Patients acceptance to have a tumor biopsy of an accessible lesion at baseline and on treatment if the lesion can be biopsied with acceptable clinical risk (as judged by the investigator).
* ECOG performance status 0 or 1.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* known history or evidence of brain metastases.
* Had surgery within the last 28 days
* Have received any non-oncology vaccine therapy used for prevention of infectious diseases including seasonal vaccinations within 28 days of study treatment.
* Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, GVAX or CRS-207
* Systemic steroids within the last 14 days
* Use more than 3 g/day of acetaminophen.
* Patients on immunosuppressive agents.
* Patients receiving growth factors within the last 14 days
* Known allergy to both penicillin and sulfa.
* Severe hypersensitivity reaction to any monoclonal antibody.
* Have artificial joints or implants that cannot be easily removed
* Have any evidence of hepatic cirrhosis or clinical or radiographic ascites.
* Have significant and/or malignant pleural effusion
* Infection with HIV or hepatitis B or C at screening
* Significant heart disease
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures
* Unable to avoid intimate contact with another individual known to be at high risk of listeriosis (e.g., newborn infant, pregnant woman, HIV-positive individual) during the course of CRS-207 treatment until completion of antibiotic regimen.
* Are pregnant or breastfeeding.
* Have rapidly progressing disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hopkins AC, Yarchoan M, Durham JN, Yusko EC, Rytlewski JA, Robins HS, Laheru DA, Le DT, Lutz ER, Jaffee EM. T cell receptor repertoire features associated with survival in immunotherapy-treated pancreatic ductal adenocarcinoma. JCI Insight. 2018 Jul 12;3(13):e122092. doi: 10.1172/jci.insight.122092. PMID 29997287

RESULTS

PARTICIPANT FLOW:
Groups:
- CY/ GVAX/ CRS-207/ Nivolumab: CRS-207: 1 × 10^9 CFU administered IV on Day 2 of Cycles 3-6
  GVAX: 5x10^8 cells administered in 6 intradermal injections on Day 2 of Cycles 1 and 2
  nivolumab: 3 mg/kg administered IV on Day 1 of Cycles 1-6
  CY: 200 mg/m^2 administered IV on Day 1 of Cycles 1 and 2
- CY/ GVAX/ CRS-207: CRS-207: 1 × 10^9 CFU administered IV Day 1 of Cycles 3-6
  GVAX: 5x10^8 cells administered in 6 intradermal injections on Day 2 of Cycles 1 and 2
  CY: 200 mg/m^2 administered IV on Day 1 of Cycles 1 and 2
Period: Overall Study
Arm/Group | CY/ GVAX/ CRS-207/ Nivolumab | CY/ GVAX/ CRS-207
Started | 51 | 42
Completed | 14 | 10
Not Completed | 37 | 32
Not completed — Progressive Disease (clinic & radio) | 35 | 24
Not completed — Death (unrelated) | 2 | 4
Not completed — Adverse Event (unrelated) | 0 | 1
Not completed — Lack of Clinical Benefit | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CY/ GVAX/ CRS-207/ Nivolumab | CY/ GVAX/ CRS-207 | Total
Number analyzed (Participants) | 51 | 42 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.08) | 63.2 (9.28) | 63.4 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 37 | 24 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 46 | 38 | 84
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 44 | 33 | 77
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS will be measured from date of randomization until death or end of followup (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis).
Time Frame: 2 years and 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
Number analyzed (Participants) | 51 | 42
months | 5.88 [4.73 to 8.64] | 6.11 [3.52 to 7.00]

2. Secondary Outcome: Number of Patients Experiencing a Grade 3 or Above Treatment-related Toxicity
Description: When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v4.03) will be counted only once for a given subject.
Time Frame: 2 years and 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
Number analyzed (Participants) | 51 | 42
Participants | 18 | 5

3. Secondary Outcome: Progression-free Survival (PFS) in Metastatic Pancreatic Cancer Patients
Description: PFS is defined as the number of months from the date of randomization to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 2 years and 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
Number analyzed (Participants) | 51 | 42
months | 2.23 [2.14 to 2.33] | 2.17 [2.00 to 2.30]

4. Secondary Outcome: Immune-related Progression-free Survival (irPFS) by IRRC in Metastatic Pancreatic Cancer Patients
Description: irPFS is defined as the number of months from the date of randomization to disease progression (PD or relapse from CR as assessed using irRC RECIST 1.1 criteria) or death due to any cause. Per irRC criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in tumor burden compared with baseline, Progressive Disease (PD) is >20% increase in tumor burden compared with nadir, Stable Disease (SD) is <30% decrease in tumor burden compared with baseline or <20% increase in tumor burden compared to nadir.
Time Frame: 2 years and 7 months
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
Number analyzed (Participants) | 51 | 42
months | 2.27 [2.17 to 2.33] | 2.23 [2.10 to 2.40]

5. Secondary Outcome: Time to Progression (TTP) by RECIST 1.1 in Metastatic Pancreatic Cancer Patients
Description: Time to progression (TTP) is defined as the time from randomization to the date of documented disease progression as defined by RECIST 1.1 criteria. Individuals are censored at the date of the last radiological assessment that occurs prior to any of the following: death, switch to another anti-cancer therapy, or end of follow-up. Individuals without follow-up or baseline measurements are censored at 1 day. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 2 years and 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
Number analyzed (Participants) | 51 | 42
months | 2.20 [2.10 to 2.33] | 2.20 [2.00 to 2.30]

6. Secondary Outcome: Number of Participants With Partial Response (PR) or Complete Response (CR) as Defined by RECIST 1.1 in Metastatic Pancreatic Cancer Patients
Description: Per RECIST 1.1 criteria, PR is defined as =>30% decrease in sum of diameters of target lesions and CR is the disappearance of all target lesions.
Time Frame: 2 years and 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
Number analyzed (Participants) | 51 | 42
Participants | 1 | 1

7. Secondary Outcome: Tumor Marker Kinetics (CA 19-9) in Patients With Baseline Abnormal Levels as Measured by Number of Participants With Stable or Responding CA19-9 Concentration
Description: Number of participants with stable or responding (<50% increase of serum CA19-9 concentration) at 120 days.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
Number analyzed (Participants) | 51 | 42
Participants | 18 | 7

ADVERSE EVENTS:
Time Frame: 2 years and 7 months
Arm/Group | Arm A: CY/ GVAX/ CRS-207/ Nivolumab | Arm B: CY/ GVAX/ CRS-207
All-Cause Mortality (participants affected / at risk) | 45/51 | 36/42
Serious Adverse Events (participants affected / at risk) | 5/51 | 1/42
Other Adverse Events (participants affected / at risk) | 46/51 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: CY/ GVAX/ CRS-207/ Nivolumab (N=51) | Arm B: CY/ GVAX/ CRS-207 (N=42)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
LISTERIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: CY/ GVAX/ CRS-207/ Nivolumab (N=51) | Arm B: CY/ GVAX/ CRS-207 (N=42)
VACCINATION SITE ERYTHEMA (General disorders) | 46 | 40
VACCINATION SITE INDURATION (General disorders) | 41 | 31
CHILLS (General disorders) | 42 | 29
VACCINATION SITE PRURITUS (General disorders) | 36 | 30
PYREXIA (General disorders) | 38 | 27
VACCINATION SITE PAIN (General disorders) | 34 | 29
VACCINATION SITE DISCOMFORT (General disorders) | 22 | 21
FATIGUE (General disorders) | 23 | 12
INFLUENZA LIKE ILLNESS (General disorders) | 13 | 8
VACCINATION SITE OEDEMA (General disorders) | 9 | 8
VACCINATION SITE SWELLING (General disorders) | 3 | 5
VACCINATION SITE VESICLES (General disorders) | 5 | 3
VACCINATION SITE REACTION (General disorders) | 5 | 2
VACCINATION SITE BRUISING (General disorders) | 4 | 2
PAIN (General disorders) | 2 | 3
NAUSEA (Gastrointestinal disorders) | 17 | 19
VOMITING (Gastrointestinal disorders) | 4 | 5
SINUS TACHYCARDIA (Cardiac disorders) | 7 | 6
TACHYCARDIA (Cardiac disorders) | 5 | 2
HEADACHE (Nervous system disorders) | 10 | 6
DIZZINESS (Nervous system disorders) | 4 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 | 2
HYPERTENSION (Vascular disorders) | 6 | 4
HYPOTENSION (Vascular disorders) | 6 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT02243371/Prot_SAP_000.pdf